CLINICAL TRIAL: NCT06068582
Title: Don't be Late! Postponing Cognitive Decline and Preventing Early Unemployment in People With Multiple Sclerosis
Acronym: DBL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Universiteit Leiden (Other); Personal Fitness Nederland (Unknown); MS Vereniging Nederland (Unknown); Merck BV (Unknown); Genzyme, a Sanofi Company (Industry); MS Sherpa (Unknown)
Responsible Party: Principal Investigator, Hanneke Hulst, Professor, Universiteit Leiden
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL82007.018.23; NWA.1292.19.064 (Other Grant/Funding Number: Dutch National Research agenda (NWA))
Record Dates: First submitted 2023-08-25; First posted 2023-10-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cognition; Exercise; Employment; Prevention; Health-related Quality of Life
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization will be done by investigators who are not involved in data collection and analyses. Intervention will be carried out by people not involved in data collection and analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Strengthening the brain (Experimental): Participants receive 30 minutes of 1-on-1 fitness training, dietary advice, and mental coaching, in addition to twice 20 minutes fitness at home, and 60 minutes of cognitive training each week for four months.
  Interventions: Behavioral: Strenghtening the brain
- Strengthening the mind (Experimental): Partiicpants receive biweekly 1-on-1 coaching by a trained work-coach who has MS to identify challenges at work and implement solutions. It is completed when satisfactory solutions have been implemented for all challenges or after four months.
  Interventions: Behavioral: Strengthening the mind
- Enhanced usual care (No Intervention): Participants receiving general information about cognitive impairment in MS and following care as usual for four months.

INTERVENTIONS:
Behavioral: Strenghtening the brain — Lifestyle intervention containing physical exercise, lifestyle coaching, and cognitive training. The programme contains weekly 30 minutes 1-on-1 fitness and lifestyle coaching with two moments of exercise at home for 20 minutes. Online computerized cognitive training will be done for 60 minutes per week.
  Arms: Strengthening the brain
Behavioral: Strengthening the mind — Work-focused intervention combining the capability approach and the participatory approach. Together with a work-coach who has been diagnosed with MS themselves, participants will assess important work values, discover challenges participants are facing, think of solutions for these challenges, develop a plan of action and implement these solutions.
  Arms: Strengthening the mind

SUMMARY:
The goal of this randomized controlled trial is to compare the effectiveness of two innovative interventions aimed at preventing cognitive decline and work-related problems to enhanced usual care in improving quality of life in people with multiple sclerosis. Secondary objectives are:

* to compare the effectiveness of the investigated interventions in improving cognitive, psychological, and work functioning, and in enhancing the brain's functional network
* to examine which factors (i.e., baseline cognitive, psychological, work, and brain MRI-parameters) are predictive of the response to the investigated interventions
* aim to qualitatively reflect on the process and outcome of the investigated interventions considering the perspectives of relevant stakeholders to allow for smooth and successful implementation in clinical practice

Participants will follow the intervention for four months, with follow-up measurements at six months after intervention and 12 months after intervention.

DETAILED DESCRIPTION:
Background Up to 65% of the people with multiple sclerosis (PwMS) develop cognitive deficits that severely affect daily life functioning and PwMS' quality of life. Moreover, approximately 65% of all patients end up unemployed within five years after diagnosis. Current treatments mostly focus on symptom management and return to work, which may be too late. It is hypothesized that timely interventions will help prevent or delay cognitive decline and work-related problems in PwMS, thereby improving quality of life.

Objectives

Primary Objective:

To compare the effectiveness of the investigated interventions with enhanced usual care in improving quality of life.

Secondary Objectives:

1. To compare the effectiveness of the investigated interventions in improving cognitive, psychological and work functioning, and in enhancing the brain's functional network.
2. To examine which factors (i.e. baseline cognitive, psychological, work and brain MRI-parameters) are predictive of the response to the investigated interventions.
3. To qualitatively reflect on the process and outcome of the investigated interventions considering the perspectives of relevant stakeholders to allow for smooth and successful implementation in clinical practice.
4. To compare the cost-effectiveness of the investigated interventions.

Material and methods A randomized controlled trial with three arms and three follow-up visits over a total time period of 16 months. During these visits researchers will gather information from questionnaires, neuropsychological examination, MRI and blood sampling. All participants (N= 240) have a confirmed MS diagnosis according to the McDonald 2017 criteria, have subclinical cognitive impairment and are aged between 18 and 67. Participants will be randomly assigned to one of the three arms (N=90 in each arm). Interviews will be conducted with 12-15 participants from both interventions, 10-12 sport coaches, 8-12 work coaches and 10-12 supervisors from the workplace.

'Strengthening the brain' (4 month-program) consists of weekly 30 minutes 1-on-1 exercise and lifestyle coaching in combination with two moments per week unsupervised exercises at home and a home-based online computerized cognitive training. 'Strengthening the mind' (4 month-program) consists of biweekly contact with work coaches who are all diagnosed with MS themselves. 'Enhanced usual care' entails an appointment with a researcher in addition to usual care.

Results The primary outcome is change in quality of life as measured with the 36-item Short Form. Several secondary outcomes will be collected: cognitive, psychological, cost-effectiveness, structural- and functional brain, neurological, physiological, and qualitative measures.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed MS diagnosis according to the McDonald 2017 criteria
* Age between 18 and 67
* No changes in disease modifying therapy prior to inclusion (i.e., no changes in last 3 months) - this criterion only applies at inclusion to ensure participants are in a stable situation at the start of the study and for follow-up measures, changes in treatment will be registered but will not result in exclusion from the study
* no current relapse or steroid treatment in the six weeks prior to study visits
* presence of mild cognitive deficits (at least one test with a Z-score of -1.0 to -1.99 below norm scores of healthy controls on the Minimal Assessment of Cognitive Function in Multiple Sclerosis (MACFIMS) battery
* being able to participate in an exercise intervention (i.e., EDSS < 6.0)
* fulfilling safety criteria for MRI (no metal inside body, not pregnant, no claustrophobia)

Exclusion Criteria:

* presence of neurological (other than MS) and psychiatric disorders
* a current or history of drug or alcohol abuse
* being unable to speak or read Dutch
* currently on sick leave for a period of 6 weeks or longer
* currently pregnant

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-04-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | Baseline, Month 4, Month 10, and Month 16
  Quality of life assessed using the 36-item Short Form. Item-scores are summed and transformed into a total score that ranges 0-100. Higher score corresponds with better quality of life.

SECONDARY OUTCOMES:
Information processing speed | Baseline, Month 4, Month 10, and Month 16
  Information processing speed is assessed using the Symbol Digit Modalities Test (SMDT). The total responses made in 90 seconds is administered. Higher amount of correct responses equals better information processing speed.
Information processing speed | Baseline, Month 4, Month 10, and Month 16
  Information processing speed is assessed using the Paced Auditory Serial Addition Test (PASAT). The total correct answers given, out of 60, is administered. Higher amount of correct responses equals better information processing speed.
Verbal fluency | Baseline, Month 4, Month 10, and Month 16
  Verbal fluency is assessed using the Dutch adaptation of the Controlled Oral Word Association Test; Dutch Letter Fluency Test. Total number of correct words will be administered. Higher score corresponds with better verbal fluency.
Spatial Processing | Baseline, Month 4, Month 10, and Month 16
  Spatial Processing is assessed using the Judgement of Line Orientation. Total correct responses, with maximum 30, will be administered. Higher score corresponds with better spatial processing.
Verbal New Learning and Memory | Baseline, Month 4, Month 10, and Month 16
  New Learning and Memory is assessed using the California Verbal Learning Test, second edition (CVLT-II). Direct recall on the CVLT-II will be administered using number of correctly remembered items over learning trials 1-5. Delayed recall on CVLT-II will be administered using number of correctly remembered items 20 minutes after learning trail 5. Maximum scores for direct recall, delayed recall, and recognition are set at 80, 16, and 44, respectively. Higher score equals better verbal learning and memory.
Visual New Learning and Memory | Baseline, Month 4, Month 10, and Month 16
  New Learning and Memory is assessed using the Brief Visuospatial Memory Test-Revised (BVMT-R). Direct recall on BVMT-R will be administered using number of correctly remembered items over learning trials 1-3. Delayed recall on BVMT-R will be administered using number of correctly remembered items 25 minutes after learning trail 3. Maximum scores for direct recall, delayed recall, and recognition are set at 36, 12, and 12, respectively. Higher score equals better visual learning and memory.
Executive Function | Baseline, Month 4, Month 10, and Month 16
  Executive Function is assessed using the Delis-Kaplan Executive Function System. Total correct sorts will be administered, with a maximum of 16 sorts. A higher score suggests better executive functioning.
Self-Reported Cognitive Functioning | Baseline, Month 4, Month 10, and Month 16
  Self-Reported Cognitive Functioning is assessed using the Multiple Sclerosis Neuropsychological Screening Questionnaire. Maximum score of 70 can be reached, with a score of 27 or higher indicating presence of neuropsychological problems.
Work Participation and Productivity | Baseline, Month 4, Month 10, and Month 16
  Work Participation and Productivity is assessed using the Work Productivity and Activity Impairment Questionnaire: General Health, which administers the effect of health-problems on ability to work. Scores are calculated as percentages, with higher numbers indicating greater impairment and less productivity.
Work Difficulties | Baseline, Month 4, Month 10, and Month 16
  Work Difficulties are assessed using the Multiple Sclerosis Work Difficulties Questionnaire. The questionnaire consists of 23 items, which can be grouped into three subscales: psychological/cognitive barriers, physical barriers, and external barriers. The maximum score of each subscale is 100, with higher scores indicating higher perceived difficulties. Total score consists of an average of the three subscale scores.
Capability to carry out Work Activities | Baseline, Month 4, Month 10, and Month 16
  Capability to carry out Work Activities is assessed using the Capability Set for Work Questionnaire. This questionnaire evaluates for seven valued work aspects whether, A) it is important to the worker, B) their work offers sufficient opportunities to do it, and C) it can be achieved, on a 5-point Likert scale.
Quality of Working Life | Baseline, Month 4, Month 10, and Month 16
  Quality of Working Life is assessed using the Quality of Working Life Questionnaire for Cancer Survivors. The questionnaire consists of five subscales: meaning of work, perception of the work situation, atmosphere in the work environment, understandings and recognition in the organisation, and problems due to health situation. The overall score and sum scores of the subscales are calculated with a standardised score 0-100. Higher score corresponds with better quality of working life.
Grey Matter Volume of the Brain | Baseline, Month 4, and Month 16
  Grey Matter Volume will be determined using FSL-SIENAX, after lesion filling on the 3DTI.
White Matter Volume of the Brain | Baseline, Month 4, and Month 16
  White Matter Volume will be determined using FSL-SIENAX, after lesion filling on the 3DTI.
Total Brain Volume | Baseline, Month 4, and Month 16
  Total Brain Volume will be determined using FSL-SIENAX, after lesion filling on the 3DTI.
Volumes of Deep Grey Matter Structures | Baseline, Month 4, and Month 16
  Volumes of Deep Grey Matter Structures will be determined using FIRST.
Cortical Thickness | Baseline, Month 4, and Month 16
  Cortical Thickness will be determined using Freesurfer.
White Matter Integrity | Baseline, Month 4, and Month 16
  White Matter Integrity will be determined using Diffusion Tensor Imaging
Functional Connectivity | Baseline, Month 4, and Month 16
  Functional Connectivity will be determined using Resting-State fMRI
Regional Functional Activation | Baseline, Month 4, and Month 16
  Regional Functional Activation will be determined using Task-Based fMRI
Fatigue | Baseline, Month 4, Month 10, and Month 16
  Fatigue will be assessed using the Checklist Individual Strength. The questionnaire consists of 20 items, scored on a 7-point Likert scale. Fatigue is a subscale of the questionnaire, and is scored by adding the scores of the items, where a higher score corresponds with more fatigue.
Mood and Anxiety | Baseline, Month 4, Month 10, and Month 16
  Mood and Anxiety will be assessed using the Hospital Anxiety and Depression Scale. The questionnaire consists of 14 items on a 4-point Likert scale. The range of scores is 0-21 where a higher score equals more complaints of anxiety and depression.
Resilience | Baseline, Month 4, Month 10, and Month 16
  Resilience will be assessed using the Connor Davidson Resilience Scale. Total score ranges 0-100, with higher scores reflecting greater resilience.
Perceived Level of Stress | Baseline, Month 4, Month 10, and Month 16
  Perceived Level of Stress will be assessed using the Perceived Stress Scale. Total score ranges 0-40, with higher scores indicating higher perceived stress.
Social Mindfulness | Baseline, Month 4, Month 10, and Month 16
  Social Mindfulness will be assessed using the SoMi paradigm by van Doesum et al. (2013). Choices that are made are scores as mindful (1) or unmindful (0). Final score will be computed by averaging the scores over all decisions, resulting in a number between 0 (unmindful) and 1 (mindful).
Social Participation | Baseline, Month 4, Month 10, and Month 16
  Social Participation will be assessed using the PROMIS 'Ability to Participate in Social Roles and Activities' item bank. The questionnaire consists of eight items that can be scored on a 5-point Likert scale. Higher scores indicate better ability to participate in social roles and activities.
MS-related disability | Baseline, Month 4, Month 10, and Month 16
  MS-related disability will be assessed using the Expanded Disability Status Scale. This scale ranges from 0.0 to 10.0, where a higher score indicates worse disability.
Balance | Baseline, Month 4, and Month 16
  Balance will be assessed using the Mini-BESTest. The test contains 14 items where a total score of 28 points can be achieved, where a score <19 induces an increased risk of falling.
Walking Speed | Baseline, Month 4, and Month 16
  Walking Speed will be assessed using the Timed 25-Foot Walk.
Endurance | Baseline, Month 4, and Month 16
  Endurance will be assessed using the Shuttle Walk Test according to the protocol of Singh et al. (1992).
Grip Strength | Baseline, Month 4, and Month 16
  Grip Strength will be assessed using a JAMAR hand-held dynamometer.
Upper Limb Dexterity | Baseline, Month 4, and Month 16
  Upper Limb Dexterity will be assessed using the 9-Hole Peg Test and the Purdue Pegboard Test.
Lost Productivity Costs | Baseline, Month 4, Month 10, and Month 16
  Lost Productivity Costs will be assessed using the iMTA Productivity Cost Questionnaire. The questionnaire consists of three modules measuring absenteeism, presenteeism, and productivity loss from unpaid work.
Societal Costs including Healthcare, Patient, and family | Baseline, Month 4, Month 10, and Month 16
  Societal Costs will be assessed using the iMTA Medical Consumption Questionnaire.
Quality Adjusted Life Years | Baseline, Month 4, Month 10, and Month 16
  Quality Adjusted Life Years will be assessed using the EuroQol five-dimensional Questionnaire. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Higher scores indicate more problems considering the dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Hanneke E Hulst, Principal Investigator — Leiden University
Locations (1):
- Amsterdam University Medical Centers, location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data relating to the main outcomes will be shared in online repository. Coded data will be published in an online scientific archive for the purpose of future research, in line with Open Science practices, and for the verification of findings. These data would not be traceable as they are not linked in any way to personal data. MRI data will be stored in OSF and other platforms that may accommodate the large capacity of the data set.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: All data will become available after the project has finished. An embargo period of one year will be used. Coded data will be published in an online scientific archive without unlimited time.
Access Criteria: Coded data that cannot be traceable to the participant identifying information will be published in an online repository

REFERENCES:
- [Derived] Aarts J, Saddal SRD, Bosmans JE, de Groot V, de Jong BA, Klein M, Ruitenberg MFL, Schaafsma FG, Schippers ECF, Schoonheim MM, Uitdehaag BMJ, van der Veen S, Waskowiak PT, Widdershoven GAM, van der Hiele K, Hulst HE; Don't be late! consortium. Don't be late! Postponing cognitive decline and preventing early unemployment in people with multiple sclerosis: a study protocol. BMC Neurol. 2024 Jan 15;24(1):28. doi: 10.1186/s12883-023-03513-y. PMID 38225561